CLINICAL TRIAL: NCT01339832
Title: Capecitabine and Oxaliplatin Prior and Concurrent to Preoperative Pelvic Radiotherapy in Patients With Locally Advanced Rectal Cancer: A Survival Analysis.
Brief Title: An Observational Study of Xeloda (Capecitabine) and Oxaliplatin Prior and Concurrent To Preoperative Pelvic Radiotherapy in Patients With Locally Advanced Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21875
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study is a follow-up study of protocol ML18280. Survival data of patients who took part in and concluded study ML18280 will be collected for up to 5 years after LPLV of ML18270.

ELIGIBILITY:
Inclusion Criteria:

* Patients who took part in and concluded study ML18280 according to protocol

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients having taken part in study ML18280
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Switzerland (5):
  - Basel
  - Chur
  - Lucerne
  - Sankt Gallen
  - Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who were treated in ML18280 base study were followed-up two, three, four years and if necessary five years after the last surgery in Switzerland (5 centers) and data concerning to the adjuvant therapy, surveillance visit, tumor recurrence or second carcinoma and survival status were collected.
Pre-assignment Details: Of the 56 participants in the ML18280 base study, 51 were included in ML21875 study. Retrospective data was documented for 14 participants and prospective data was obtained for 37 participants.
Groups:
- Overall: Participants with histologically proven local advanced T3/T4 rectal carcinoma with or without nodal involvement who had participated in study ML18280 were enrolled and no active treatment was given during this study
Period: Overall Study
Arm/Group | Overall
Started | 51
Completed | 37
Not Completed | 14
Not completed — Lost to Follow-up | 3
Not completed — Death | 11

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all the participants who fulfilled the inclusion criteria for this study. This population includes participants who gave informed consent and also those who died or were lost to follow-up before start of ML21875 study.
Arm/Group | Overall
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression free survival (PFS) was measured from the date of first administration of study medication in ML18280 study to the date of progression or death, whatever the cause. In participants with measurable disease, progression was defined according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.0. Participants with neither tumor recurrence nor death were censored at the last tumor assessment date they were known to have not progressed (last date of diagnostic procedure or diagnostic marker reported in the surveillance). PFS time in days was calculated as PFS [days]= date of tumor recurrence/death date of first intake + 1, if participant had tumor recurrence confirmed by diagnostic imaging or participant died, then PFS [days] =last diagnostic procedure/marker date- date of first intake+ 1, and if participant survived without tumor recurrence PFS time in months was calculated as PFS [months]= 12 * PFS [days] /365.25
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (Full Range); unit: months
Arm/Group | Overall
Number analyzed (Participants) | 51
months | 15.4 [7.3 to 60.0]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as time from date of first administration of the study medication in ML18280 study to date of death from any cause. Participants without documented date of death were assumed to be alive and were censored at the latest of the following dates: last date alive on survival status pages, last date known to be alive on survival status pages, and last date of tumor assessment (diagnostic procedures or markers) on surveillance pages. OS time in days was calculated as OS [days] =date of death date of first intake+ 1, for participants who died, OS [days]= censoring date date of first intake+ 1, for participants alive, and OS time in months was calculated as OS [months]= 12 *OS [days] /365.25
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (Full Range); unit: months
Arm/Group | Overall
Number analyzed (Participants) | 51
months | 22.51 [10.3 to 60.0]

3. Secondary Outcome: Tumor Recurrence Rate (Local and Distant)
Description: Participant with tumor recurrence were determined by the presence or absence of date of tumor recurrence detection. In case of absence of empty tumor recurrence date it was considered that the participant had not experienced tumor recurrence. Participants with local tumor recurrence ('Was it local to the primary tumor?' answered 'yes'.) compared to participants with distant tumor recurrence (specification for other tumor location given).
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 51
participants
  Participants with Tumor Recurrence | 16
  Participants with Tumor Recurrence- Local | 4
  Participants with Tumor Recurrence- Distant | 12

4. Secondary Outcome: Type of Adjuvant Chemotherapy
Description: The type of therapies administered after primary treatments (chemotherapy, surgery or radiation) was reported
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 51
participants
  Folfox | 2
  Xelox | 10
  Xeloda mono or 5-FU mono | 14
  Other (Biologics) | 2
  Xeloda + Irinotecan | 2
  No adjuvant chemotherapy | 21

5. Secondary Outcome: Length of Adjuvant Chemotherapy
Description: The length of adjuvant chemotherapy was defined as time between first start date to last stop date of adjuvant chemotherapy regimen. Length of adjuvant chemotherapy was calculated as length [days] = last stop date - first start date + 1, missing day of start and stop date was replaced by 1.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (Full Range); unit: days
Arm/Group | Overall
Number analyzed (Participants) | 51
days | 49.0 [0 to 1149]

6. Secondary Outcome: Compliance to Diagnostic Procedures in Surveillance
Description: The surveillance compliance was calculated per participant in percent and frequencies for methods of diagnostic procedure adhered to, taking into account all expected procedures in the time span the participant participated and was based on the Swiss Society of Gastroenterology (SGG) follow-up care recommendations
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 51
participants
  X-ray Chest | 32
  Colonoscopy | 40
  Computed Tomography (CT) | 61
  Endosonography | 30
  Magnetic resonance imaging | 14
  Unknown | 1
  Balloon Dilatation (BD) Ileostoma | 1
  BD Ileostoma+ Oesophagus-Gastroduodenum | 1
  Colon monocontrast | 1
  Colonoscopy Polypectomy | 1
  CT Abdomen | 1
  CT Thorax + Abdomen | 1
  Densitometry | 1
  Duplex Sonography | 1
  Enteroscopy | 1
  Ergometry | 1
  Oesophagus-gastroduodenoscopy | 4
  Fine Needle Puncture Lung | 1
  Gastroduodenoscopy | 3
  Gastrophinpassage | 1
  Gastroscopy | 1
  Ileocoloscopy | 2
  Ileoscopy | 1
  X-ray Lumbar Spine | 1
  Manometry | 2
  X-ray Pelvis | 1
  Positron emission tomography (PET) | 1
  PET-CT | 11
  Proctoscopy | 2
  Rectoproctoscopy | 3
  Rectoscopy | 7
  Rectosigmoidoscopy | 4
  Scintigraphy | 1
  Scintigraphy Lung | 1
  Sigmoidoscopy | 2
  Sonography | 6
  Starre Rectoscopy | 1
  Scintigraphy Bone Scan | 1
  Ultrasound | 6
  Ultrasound Abdomen | 5
  Video Bronchoscopy | 1
  X-ray Abdomen | 3
  X-ray Barium Swallow | 1
  X-ray Spine | 1

7. Secondary Outcome: Long Term Side Effects
Description: Long term side effects for bowel and urinary function was assessed. Bowel function was assessed in terms of mean bowel frequency, regular use of constipating agents as well as fecal incontinence. Urinary function was evaluated according to the presence (YES or NO) of incontinence. Overall participant satisfaction was assessed in terms of satisfaction with bowel, stoma and urinary function on a 4-stage scale (very good, good, poor, and very poor). In case of different assessment(s) of bowel or urinary function within the same surveillance period, the assessment with worst grade was documented and reported.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 51
participants
  Bowel frequency, <3 | 13
  Bowel frequency, 3-5 | 8
  Bowel frequency, 6-9 | 5
  Bowel frequency, >9 | 1
  Use of constipating agents | 16
  Fecal incontinence | 17
  Urinary incontinence | 2
  Overall participant satisfaction, very good | 2
  Overall participant satisfaction, good | 10
  Overall participant satisfaction, poor | 8
  Overall participant satisfaction, very poor | 6

8. Secondary Outcome: Incidence of Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 51
participants
  Number of participants with AE | 4
  Number of participants with SAE | 1

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 1/51
Other Adverse Events (participants affected / at risk) | 3/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=51)
Polyneuropathy (Nervous system disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=51)
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Hypersensitivity (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.